CLINICAL TRIAL: NCT05576402
Title: Endoscopic Scoring System Utilization for Inflammatory Bowel Disease Activity Assessment
Brief Title: Endoscopic Scoring System Utilization in Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno (Other)
Responsible Party: Principal Investigator, Juan Lasa, Principal investigator, Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno
Other Study IDs: 333
Record Dates: First submitted 2022-10-08; First posted 2022-10-12 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: colonoscopy — endoscopic exploration of colonic mucosa to evaluate inflammatory activity in patients with either Crohn's disease or ulcerative colitis
  Other Names: endoscopic score assessment

SUMMARY:
Inflammatory bowel diseases comprise two distinctive entities: Crohn's disease and ulcerative colitis. During the last decade, endoscopic assessment of inflammation has become relevant since it is a prognostic factor. As a consequence, therapeutic targets now contemplate mucosal healing as part of the goals to be achieved. Endoscopic scores for Crohn's disease and ulcerative colitis have been developed to objectively assess the mucosal inflammatory activity. Although they may have some limitations, these scores have been widely accepted in referral centers, especially since they have been adopted as standard evaluation in inflammatory bowel disease clinical trials . However, their use in the setting of endoscopic practice outside centers with a high volume or with less experience in clinical trials is not known.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent colonoscopy for the evaluation of mucosal inflammatory activity
* Patients with an established diagnosis of either Crohn's disease or ulcerative colitis

Exclusion Criteria:

* Sigmoidoscopies performed in ulcerative colitis for the assessment of mucosal inflammatory activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have already received a diagnosis of either Crohn's disease or ulcerative colitis
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Endoscopic score report | January 2018-October 2022
  Proportion of colonoscopy reports among inflammatory bowel disease patients which include an endoscopic score to assess inflammatory activity

CONTACTS AND LOCATIONS:
Overall Officials: Juan S Lasa, MD, Principal Investigator — Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno
Locations (1):
- CEMIC, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No